CLINICAL TRIAL: NCT03565159
Title: Pneumococcal Vaccination to Accelerate Immune Recovery in Sepsis Survivors
Acronym: VACIRiSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 430321; 2017-002236-17 (EudraCT Number)
Record Dates: First submitted 2018-05-25; First posted 2018-06-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — 13-valent pneumococcal vaccine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomised 1:1 to receive one single 0.5ml dose of active or placebo Investigational Medicinal Product at baseline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevenar 13 (Active Comparator): A volume of 0.5ml will be drawn up into a syringe and labelled with an Annex 13 label.
  Interventions: Biological: Prevenar 13
- Sodium chloride 0.9% (Placebo Comparator): A volume of 0.5ml will be drawn up into a syringe and labelled with an Annex 13 label.
  Interventions: Other: Sodium Chloride 0.9%

INTERVENTIONS:
Biological: Prevenar 13 — Pneumococcal polysaccharide conjugate vaccine
  Arms: Prevenar 13
Other: Sodium Chloride 0.9% — Placebo
  Arms: Sodium chloride 0.9%

SUMMARY:
The VACIRiSS trial is a phase-IV, multi-centre placebo controlled randomised trial of conjugate pneumococcal vaccine in adult sepsis survivors.

DETAILED DESCRIPTION:
The aim of VACIRiSS trial is to evaluate the immunogenicity and heterologous effects of single dose 13-valent conjugate pneumococcal vaccine (PCV-13) in preventing infection related rehospitalisation in sepsis survivors and to collect outcome event data with necessary precision to inform future definitive trial design.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following inclusion criteria are eligible to participate in the trial.

* Male or female adult patients aged 18 years or older on the date of screening for the trial
* Registered with a General Practitioner
* Reason for admission to intensive care unit or high dependence unit (HDU) was sepsis
* Clinical condition has improved and the patient is ready for step down to HDU or ward based care in the next 24 - 48 hours
* Provision of written informed consent by the patient OR by patient's Legal Representative OR Professional Consultee.

Exclusion Criteria:

Patients who meet one or more of the following will be excluded from the trial.

* Core temperature ≥38.0°C within the past 24 hours prior to study IMP administration. As with other vaccines, the administration of Prevenar 13 should be postponed in subjects suffering from acute, severe febrile illness. However, the presence of a minor infection, such as a cold, should not result in the deferral of vaccination.
* Hypersensitivity reaction (e.g., anaphylaxis) to any component of Prevenar 13 or any diphtheria toxoid-containing vaccine.
* Recent vaccination defined as any vaccination administered to subjects within 7 days of enrolment.
* Pregnant and lactating women.
* Limitations of care set including not for resuscitation, not for readmission to critical care.
* Residence in a nursing home, long-term care facility, or other institution, or requirement of semiskilled nursing care. (An ambulatory subject who was a resident of a retirement home or village is eligible for the trial.)
* As the IMP is administered intra muscularly, coagulopathy defined as platelet count less than 50 x 109/L and/or International Normalized Ratio (INR) greater than 1.3. For this exclusion criteria bloods taken within 72 hours of screening are valid. If these standard of care blood results are not available, then these should form part of the screening bloods for assessing eligibility.
* Splenectomy (previous or in the current admission)
* Diagnosis of pneumococcal sepsis in the current admission
* APACHE II score defined Immune deficiency or suppression, defined as presence of 1 or more of the following conditions:
* Documented human immunodeficiency virus (HIV) infection at any time-point pre-trial. If previous results are not available and/or current admission is not due to HIV infection, these patients do not need new testing and are considered eligible for the trial.
* leukaemia (presence defined as having been treated by or been eligible for treatment by radiotherapy and/or chemotherapy within the last 5 years)
* lymphoma (presence defined as having been treated by or been eligible for treatment by radiotherapy and/or chemotherapy within the last 5 years) Hodgkin disease (presence defined as having been treated by or been eligible for treatment by radiotherapy and/or chemotherapy within the last 5 years)
* multiple myeloma (presence defined as having been treated by or been eligible for treatment by radiotherapy and/or chemotherapy within the last 5 years)
* malignancy (defined as presence of any malignancy that had been treated by or had been eligible for treatment by radiotherapy and/or chemotherapy within the last 5 years)
* chronic renal failure (defined as receipt of renal dialysis or transplant) or nephrotic syndrome
* receipt of immunosuppressive therapy, including steroids, within 3 months of study vaccine administration (For corticosteroids, prednisone or equivalent 0.5 mg/kg/day for 14 days or longer. Inhaled, intra- articular, and topical steroids are not considered immunosuppressive).
* Receipt of an organ or bone marrow transplant with ongoing immunosuppressive medications. Failed previous transplant patients not currently on immunosuppression are eligible.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Primary - Time to Event | Up to 365 days
  Comparison of the time taken for infection related rehospitalisation or death between intervention and control arms.

SECONDARY OUTCOMES:
Secondary - Precision Estimates | Up to 365 days
  Outcome event data to inform future definitive trial, including:
  - proportion of rehospitalisation
Secondary - Precision Estimates | Up to 365 days
  - proportions of reinfections
Secondary - Precision Estimates | Up to 365 days
  - proportions of reinfection related rehospitalisation
Secondary - Precision Estimates | Up to 365 days
  - time to first all cause rehospitalisation and
Secondary - Precision Estimates | Up to 365 days
  - time to first infection requiring antibiotic therapy

OTHER OUTCOMES:
Exploratory - Immune recovery patterns | Day 0 (baseline) to Day 90
  Differences between the intervention and control arms of the following:
  anti-pneumococcal antibody
Exploratory - Immune recovery patterns | Day 0 (baseline) to Day 90
  Differences between the intervention and control arms of the following:
  B cell subsets, T cell subsets and monocyte HLA-DR and PD-1 expression), function and leukocyte transcriptome

CONTACTS AND LOCATIONS:
Overall Officials: Manu Shankar-Hari, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust and King's College London
Locations (12):
- United Kingdom (12):
  - Belfast Health and Social Care Trust, Belfast
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Lothian, Edinburgh
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Aneurin Bevan University Health Board, Newport
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Undecided
Access Criteria: Undecided